CLINICAL TRIAL: NCT06380868
Title: Intravascular Imaging-guided Versus Angiography-guided PCI in Patients With Diabetes Mellitus: the Muticenter, Randomized, Prospective IVI-DIABETES Trial
Brief Title: IVI-guided Versus Angiography-guided PCI in Patients With Diabetes Mellitus
Acronym: IVI-DIABETES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: Shanxi Provincial People's Hospital (Other Government)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Professor, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Nanjing-2
Record Dates: First submitted 2024-03-25; First posted 2024-04-24 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Patients will undergo 1:1 randomization to either intravascular imaging (including intravascular ultrasound or optical coherence tomography)-guided DES implantation which will be the treatment group or Angio-guided DES implantation which will be the control group, stratified by research sites.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization will be performed in the catheter laboratory by an invasive nurse. Staff in the catheter laboratory will be not blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular imaging-guided PCI group (Experimental): For patients in this group, intravascular imaging will be encouraged to performed prior-to and post-coronary intervention using new generation drug-eluting stents
  Interventions: Procedure: Intravascular imaging-guided PCI
- Angiography-guided PCI group (Active Comparator): For patients in this group, implantation of a new generation drug-eluting stent will be guided by angiography only. Unless coronary artery lesion is complex or ambiguous, intravascular imaging is not allowed to be used. If intravascular imaging is used because of the reason mentioned above, post-stenting assessment is absolutely not allowed.
  Interventions: Procedure: Angiography-guided PCI group

INTERVENTIONS:
Procedure: Intravascular imaging-guided PCI — Intravascular imaging including intravascular ultrasound or optical coherence tomography.
  Arms: Intravascular imaging-guided PCI group
Procedure: Angiography-guided PCI group — Deployment of a drug-eluting stent under angiography.
  Arms: Angiography-guided PCI group

SUMMARY:
Intravascular ultrasound (IVUS) serves as a beneficial instrument during percutaneous coronary intervention (PCI) procedures, affording insight into lesion characteristics and stent implantation. The ULTIMATE trial recently evidenced that IVUS-guided Drug-Eluting Stent (DES) implantation notably ameliorated clinical outcomes in all-comers, especially in patients who underwent an optimal procedure defined by IVUS, as opposed to angiography guidance, resonating with findings from the IVUS-XPL study, OCTOBER trial, and RENOVATE COMPLEX PCI trial, further confirmed by more recent IVUS-ACS trial.

Optical coherence tomography (OCT) has a resolution 10 times higher than that of IVUS and can provide valuable information at each step of PCI.

Regrettably, a dearth of prospective, randomized, multicenter trials exists that scrutinize the benefits of IVI-guided as opposed to angiography-guided PCI in patients suffering from diabetes mellitus. However, several trials have presented subgroup analyses reporting the reduction of clinical events by IVUS but not OCT guidance in patients with diabetes mellitus, which served as the foundation for the design of this trial.

DETAILED DESCRIPTION:
The current study hypothesizes that IVI-guided PCI will be superior with respect to target vessel failure (TVF), including cardiac death, target-vessel myocardial infarction (TVMI), or clinically-driven TVR when compared with angiography-guided PCI in patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 ~ 80 years old,
2. Confirmed diabetes mellitus
3. Indications for undergoing percutaneous coronary intervention using a drug-eluting stent (Invasive or quantitative fractional flow reserve (QFR or FFR) <0.80)
4. Silent angina, stable angina, unstable angina, or Non-ST-elevation myocardial infarction

Exclusion Criteria:

1. Cardiogenic shock
2. Previous coronary artery bypass graft (CABG)
3. Left ventricular ejection fraction < 30%
4. Requiring oral anticoagulation medications
5. Any planned surgery within 12 months
6. Severe chronic kidney disease defined as an estimated glomerular filtration rate (eGFR) < 20 ml/min/1.73m2
7. Platelet count < 100,000 mm3
8. Contraindication to study medications or metal
9. Women of childbearing potential
10. Life expectancy < 1 year
11. Any condition likely to interfere with study processes including medication compliance or follow-up visits (e.g. dementia, alcohol abuse, severe frailty, long distance to travel for follow-up visits, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1332 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Rate of target vessel failure (TVF) | At one-year since interventions
  TVF is defined as a composite of cardiac death, target-vessel myocardial infraction, or clinically driven target vessel revascularization

SECONDARY OUTCOMES:
Rate of target vessel failure without procedure-related MI | At one-year since interventions
  Procedural-related myocardial infarction (PMI) would be excluded from the calculation of TVF
Rate of cardiac death | At one-year since interventions
  Any death without clear reasons
Rate of all-cause death | At one-year since interventions
  Any death occurs within one-year follow-up
Rate of procedure-related myocardial infarction (PMI) | Within 48 h since coronary intervention
  48 hours after coronary intervention
Rate of spontaneous myocardial infarction (SMI) | Within one-year follow-up
  MI happens between 48 h and one-year since coronary intervention
Rate of clinically-driven revascularization | At one-year since coronary artery intervention
  Target vessel revascularization was defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel was defined as the entire major coronary vessel proximal and distal to the target lesion, which included upstream and downstream branches and the target lesion itself.
Rate of stent thrombosis | At one-year since coronary artery intervention
  Definite or probable stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Jing Kan, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University, and Shan'Xi Provincial People's Hospital, China
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao XF, Kan J, Wu HY, Chen J, Chen X, Wen SY, Gong YT, Tong Q, Luo J, Shao YB, Gill BUA, Malik FTN, Santoso T, Daggubati R, Rodriguez AE, Francesco L, Rahman A, Sheiban I, Kedev S, Munawar M, Kwan TW, Wang Y, Ye F, Zhang JJ, Shou XL, Chen SL; IVI-DIABETES investigators. Intravascular imaging-guided versus angiography-guided percutaneous coronary intervention in patients with diabetes mellitus: Rationale and design of an international, multicenter, randomized IVI-DIABETES trial. Am Heart J. 2025 May;283:81-88. doi: 10.1016/j.ahj.2025.01.017. Epub 2025 Feb 4. PMID 39914556